CLINICAL TRIAL: NCT04021186
Title: An Optimization in the Postoperative Treatment in Head and Neck--surgical Patients -- Improvement in Glycemic Control to Reduce the Incidence of Hyperglycaemia and Associated Complications.
Brief Title: An Optimization in the Postoperative Treatment in Head and Neck--surgical Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associated Professor, MD, MPA, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DM-HHC
Record Dates: First submitted 2019-07-05; First posted 2019-07-16 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Hyperglycemia Steroid-induced; Hyperglycemia Stress; Surgery--Complications

STUDY DESIGN:
Intervention Model Description: Prevention of hyperglycemia. The study will involve an intervention and a control group - only the intervention group will receive different treatment and the other standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Insulin treatment using standard measurements.
  Interventions: Other: Prevention of hyperglycemia
- Control (No Intervention): Standard care.

INTERVENTIONS:
Other: Prevention of hyperglycemia — Bigger focus on postoperative blood-glucose levels in order to reduce incidents of hyperglycemia and other surgical complications.
  Arms: Intervention

SUMMARY:
Based on glycemic load (overall increase in blood glucose), it is investigated whether better glycemic control (large fluctuations in blood glucose to abnormal values are attempted) can improve the postoperative phase of head and neck surgical patients who receive Dexamethasone (glucocorticoid). Furthermore it is examined whether this optimization in treatment can result in reduced hospitalization time and fewer re-admissions.

Hypothesis:

Continuous blood glucose measurement and insulin therapy will optimize the postoperative phase of the embedded head and neck patient receiving Dexamethasone by reducing the incidence of hyperglycaemia and associated complications.

DETAILED DESCRIPTION:
After surgical intervention, an insulin resistance condition will occur because of the following stress response. This condition will for the majority of cases results in poor glycemic control - and there will be a risk of hyperglycaemia in the hospitalized patient. This condition affects all cells in the body and therefore has associated complications such as bigger risk at multiple infections, longer healingprocess, poorer fluid balance, etc. Hyperglycaemia is associated with a poorer outcome for the patient, which can cause an increase in hospitalization days and multiple re-admissions. It is also common for the postoperative patient to experience nausea and pain as a result of both surgery and anesthesia and immobilization. To counter this, the patient receives Dexamethasone (steroid treatment).

This experiment is based on the fact that there is still insufficient attention at this postoperative insulin resistance. In a large randomized study from 2001(Van den Berghe), insulin therapy was initiated for intensive patients. This study points out that even moderate increases in blood glucose are associated with increased morbidity and that insulin therapy is both capable of reducing mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* All embedded head and neck-surgical patients receiving large packs of pre-medication, including 8-16 mg glucocorticoid.
* >18 yrs.
* Expected admission time of a minimum of 1 day

Exclusion Criteria:

* Patients who do not understand and / or speak Danish
* Patients who are demented
* Patients included in primary robot surgery
* Ear-surgical patients
* Sinus surgery patients
* Day surgery patients
* Plastic surgical patients
* Patients who are scheduled to transfer to ICU
* Patients with Diabetes Mellitus type I
* Patients on dialysis
* If all preoperative blood samples and tests are not completed
* Type 2 diabetics in insulin therapy
* Anesthesia patients
* Patients who have received large packages of pre-medication twice - eg. due to cancelled operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-08-17 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Glycemic load (mmol) | 1-5 days
  All blood glucose levels of the participants will be measured every 30. min - all values will be used to make an area under the curve in final statistics.

SECONDARY OUTCOMES:
Temperature (degree celcius) | 1-5 days
  The temperature will be measured 3 times a day for each participant
C-Peptide | 1-5 days
  Blood sample - Will be measured 3 times
Strength of Hand grip (kg) | 20 days
  Will be measured 3 times. Maximal values of 3 attempts
Number of re-Hospitalizations | 30 days postoperatively
  counted
Number of re-Hospitalizations | Up to 3 months after the first discharge
  counted
Intracellular hydration (liters) | 20 days
  Will be measured by bioimpedance and blood sample of hematocrit
C-reactive protein (CRP) concentration | 20 days
  Blood sample - will be measured 3 times
Blood glucose (mmol/l) | 1-5 days - every 30. min.
  Will be measured by electronical device called Freestyle Libre (CGM)
Functional recovery | 20 days
  Performa status and FOIS (Functional Oral Intake Scale = degree of swallowing problems/dysphagia) scale will be used (points 1-7)

CONTACTS AND LOCATIONS:
Overall Officials: Jens R. Andersen, AP, MD, MPA, Principal Investigator — University of Copenhagen
Locations (1):
- Clinic for Ear, Nose and Throat Surgery, Rigshospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen SK, Olsen JQ, Jalili M, Wessel I, Andersen JR. Postoperative glycemic control in head and neck surgery. Clin Nutr ESPEN. 2025 Aug;68:691-698. doi: 10.1016/j.clnesp.2025.06.024. Epub 2025 Jun 13. PMID 40518009